CLINICAL TRIAL: NCT05857124
Title: A Pilot Study Evaluating the Efficacy of the Vielight Neuro RX Gamma in the Treatment of Post COVID-19 Cognitive Impairment
Brief Title: A Study Evaluating the Efficacy of the Vielight Neuro RX Gamma in the Treatment of Post COVID-19 Cognitive Impairment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vielight Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: VL-2023-PostCOVID-Pilot
Record Dates: First submitted 2023-05-10; First posted 2023-05-12 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Post COVID-19 Cognitive Impairment

STUDY DESIGN:
Intervention Model Description: This trial utilizes a completely remote and virtual design. It is a double blind randomized controlled trial that is expected to involve 36 participants who are confirmed to have Post- COVID cognitive impairment.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Active treatment devices (Experimental): Vielight Neuro RX Gamma active device
  Interventions: Device: Vielight Neuro RX Gamma active device
- Sham devices (Sham Comparator): Vielight Neuro RX Gamma sham device
  Interventions: Device: Vielight Neuro RX Gamma sham device

INTERVENTIONS:
Device: Vielight Neuro RX Gamma active device — The Vielight Neuro RX Gamma active device is a home-use photobiomodulation (PBM) device designed to deliver near-infrared (810 nm) light (or photons) to the brain/scalp and nasal tissues.
  Arms: Active treatment devices
Device: Vielight Neuro RX Gamma sham device — The Vielight Neuro RX Gamma sham device is a home-use device similar to the Vielight Neuro RX Gamma active device, but acting as a sham.
  Arms: Sham devices

SUMMARY:
Some people who have been infected with the virus that causes COVID-19 can experience long-term effects from their infection, known as post COVID-19 conditions (PCC) or long COVID1. The medical circles often describe it as post-acute sequelae of Covid-19 (PASC). People with post-COVID conditions can have a wide range of symptoms that can last more than four weeks or even months after infection. Sometimes the symptoms can even go away or come back again. The Centers for Disease and Prevention (CDC) listed a constellation of 19 symptoms related to post COVID-19.

In research, brain fog is prominent among the most reported neurological symptoms which also include, numbness, tingling, headache, dizziness, blurred vision, tinnitus, and fatigue that last more than a year post-infection.

Vielight Inc. has developed a compact and portable device named the "Vielight RX Gamma", which is suitable for home use. The intervention is based on the science of photobiomodulation (PBM) which utilizes certain light energy to modify cellular functions. The fundamental mechanisms of PBM are based on the absorption of photons by the mitochondria to modulate cellular functions. The Vielight Neuro RX Gamma delivers light of specific wavelengths (810 nm), power and duration to the brain/nasal cavity to achieve this. The biological process involves numerous interacting mechanisms that modulate bodily functions. One result of PBM is the benefits it could offer the post COVID-19 (long COVID) population. The Vielight Neuro RX Gamma emitting NIR might reduce inflammatory markers relevant to COVID-19 and since it pulses at 40 Hz can activate the non-inflammatory M2-genotype microglia to remove markers of Alzheimer disease, such as beta-amyloid and possibly tau deposits. Using Vielight Neuro RX Gamma, the same activation of non-inflammatory markers might occur with post COVID-19 (long-COVID) patient population as well as the reduction in the brain fog.

This trial utilizes a completely remote and virtual design. It is a double blind randomized controlled trial that is expected to involve 36 participants who are confirmed to have Post- COVID cognitive impairment. Eighteen of the participants will be randomized to the active Vielight RX Gamma protocol, and the other eighteen participants will be randomized to the sham Vielight RX Gamma regimen. The trial will study patients over 120 days and ask them to track their symptoms in a daily survey.

ELIGIBILITY:
Inclusion Criteria:

* Male or female age 18-65.
* Diagnosed with Post COVID cognitive impairment who meets WHO-defined post-COVID-19 condition
* Mini Mental State Examination (MMSE) score of <27
* Capable of filling out an online patient diary in English.

Exclusion Criteria:

* Current symptoms are explained by a psychiatric or neurological disorder
* Having or history of any major neurological or psychiatric illness
* Pregnant
* Physical, cognitive, or language impairments sufficient to adversely affect data derived from cognitive assessments or History of mild traumatic brain injury (TBI)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2025-01-16 (Actual)

PRIMARY OUTCOMES:
The change in the combined results of 7 Creyos items: Spatial Planning, Monkey Ladder, Rotations, Feature Match, Paired Associates, Token Search, Polygons. | from baseline to Day 56

SECONDARY OUTCOMES:
Creyos scores of the 5 remaining tests (i.e. Grammatical Reasoning, Spatial Span, Digit Span, Odd One Out, Double Trouble) | 0, 14, 28, 56 and 84 days
EQ-5D-5L Quality of Life | 0, 14, 28, 56 and 84 Days
Fatigue Assessment Scale (FAS) | 0, 56 and 84 Days
The perceived deficits questionnaire - 20 item version (PDQ-20) | 0, 56 and 84 days
Compliance and Technical Complications | 0 to Day 56
Modified Symptom Burden Questionnaire | 0 and 56 Days
  (Breathing Pain Fatigue Memory, Thinking and Communication Sleep Ears, Nose and Throat Stomach and Digestion Other Symptoms)

OTHER OUTCOMES:
Exploratory Endpoints | 0 to Day 56
  Statistical analysis of the Creyos changes between treatment groups may warrant further exploration of the primary endpoint model

CONTACTS AND LOCATIONS:
Locations (1):
- Ascada Research, Fullerton, California, United States

IPD SHARING:
Plan to Share IPD: No